CLINICAL TRIAL: NCT05753644
Title: The Effect of Preoperative Stellate Ganglion Block on Postoperative Atrial Fibrillation After Video-assisted Thoracoscopic Surgeries: A Randomized Controlled Trial
Brief Title: The Effect of Preoperative SGB on POAF After VATS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Juhui, professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SGB and POAF
Record Dates: First submitted 2023-02-12; First posted 2023-03-03 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation
Keywords: Postoperative atrial fibrillation; stellate ganglion block
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ropivacaine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGB group (Experimental): The subjects will accept ultrasound guided SGB in the right side of the neck in a supine position. The drug is 5 ml of 0.5% ropivacaine.
  Interventions: Procedure: stellate ganglion blocks; Drug: Ropivacaine
- control group (Placebo Comparator): The subjects will accept sham block in the right side of the neck in a supine position. A sham block is performed by subcutaneous infiltration (1 mL1% lidocaine) on the site.
  Interventions: Procedure: stellate ganglion blocks; Drug: Sham treatment

INTERVENTIONS:
Procedure: stellate ganglion blocks — At the level between C6 and C7, a 25-gauge needle is inserted laterally, and the needle tip is placed posterior to the carotid artery and anterior to the longus colli muscle using an in-plane approach.
Drug: Ropivacaine — 5 mL of 0.5% ropivacaine injected in the plane of the right stellate ganglion
  Other Names: SGB group
  Arms: SGB group
Drug: Sham treatment — 5 mL of saline injected in the plane of the right stellate ganglion
  Other Names: Control group
  Arms: control group

SUMMARY:
The aim of this study is to test if stellate ganglion block can decrease the incidence of atrial fibrillation after video-assisted thoracoscopic surgery and the way it works.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF) is a common complication after video-assisted thoracoscopic surgeries. It leads to early postoperative complications, prolonged ICU stay and hospital stay, increased hospital expense and medical system burden. POAF is hard to predict and difficult to treat. The potential mechanism of POAF is not fully understood. Since early 2020, covid-19 overwhelmed globally. Chest X-rays and CT scans prescribed enormously due to screening for covid-19 infection. Lung nodules are frequently discovered and the number of video-assisted thoracoscopic procedures is surged. Prevention and new targets of treatment of POAF need to be investigated urgently. This is a double blinded, randomized controlled trial, investigating the effect of autonomic nervous system modulation on POAF. In current study, patients with one or more POAF risks, who undergo video-assisted thoracoscopic lobectomy will be enrolled and randomized into two groups. Participants in the SGB group receive stellate ganglion blocks (SGB) preoperatively, while those in the control group receive sham blocks. All the patients receive standardized anesthesia and video-assisted thoracoscopic procedures. All of participants will be monitored with portable ECG monitoring for 48 hours to detect any POAF occurrence. Cytokines including IL-2, IL-6 and inflammatory bio-markers including C-reactive protein and white blood cell count are measured before surgery, 24h and 48h after surgery. The primary outcome is the occurrence of POAF and its duration. The sample size is calculated as 191 patients per group. The presumed result will be that SGB will lower the POAF incidence and shorten the duration after video-assisted thoracoscopic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* 1.patients undergoing elective thoracoscopic lobectomy;
* 2.patients with one or more risk factors of POAF. According to literature, risks factors of POAF including male, aged over 65, obesity (BMI>30kg/m2), cardiac co-morbidity ( hypertension, myocardial infarction, heart failure, arrhythmia, history of valve procedure), diabetes, chronic renal insufficiency (increased creatinine level), obstructive sleep apnea syndrome (diagnosed or STOP-BANG scores ≥3).

Exclusion Criteria:

* 1. patients with permanent atrial fibrillation, left ventricular or right ventricular pacemaker implantation or removal;
* 2. patients use antiarrhythmic drugs (except beta-blockers);
* 3.patients use immunosuppressive drugs preoperatively;
* 4.patients with active infection or sepsis;
* 5. patients with neurologic disorder;
* 6.patients with immune deficiency syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome is the incidence of POAF using dynamic electrocardiogram. | within 48 hours post-surgery
  Percentage of subjects who experience POAF.

SECONDARY OUTCOMES:
Secondary outcome is the level of inflammatory mediators including IL-2, IL-6, CRP, WBC count. | T0: pre-induction; T1: immediate after surgery; T2: 24 hours after T1; T3: 48 hours after T1. A cycle is 24 hours.
  The level of inflammatory mediators.

OTHER OUTCOMES:
The third outcome is the effect of stellate nerve block on postoperative analgesia using dosage of analgesic. | T1: immediate after surgery; T2: 24 hours after T1; T3: 48 hours after T1; T4: 72 hours after T1. A cycle is 24 hours.
  The effect of postoperative analgesia.
The fourth outcome is the effect of stellate nerve block on postoperative analgesia using NRSS score. | T1: immediate after surgery; T2: 24 hours after T1; T3: 48 hours after T1; T4: 72 hours after T1. A cycle is 24 hours.
  The effect of postoperative analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Ju, Principal Investigator — Peking University People's Hospital, Beijing, China
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang H, Wang Z, Zhou M, Chen J, Yao F, Zhao L, He B. Postoperative atrial fibrillation in pneumonectomy for primary lung cancer. J Thorac Dis. 2021 Feb;13(2):789-802. doi: 10.21037/jtd-20-1717. PMID 33717552
- [Result] Auer J, Weber T, Berent R, Ng CK, Lamm G, Eber B. Risk factors of postoperative atrial fibrillation after cardiac surgery. J Card Surg. 2005 Sep-Oct;20(5):425-31. doi: 10.1111/j.1540-8191.2005.2004123.x. PMID 16153272
- [Result] Koch CG, Li L, Van Wagoner DR, Duncan AI, Gillinov AM, Blackstone EH. Red cell transfusion is associated with an increased risk for postoperative atrial fibrillation. Ann Thorac Surg. 2006 Nov;82(5):1747-56. doi: 10.1016/j.athoracsur.2006.05.045. PMID 17062241
- [Result] Vidotti E, Vidotti LFK, Arruda Tavares CAG, Ferraz EDZ, Oliveira V, de Andrade AG, Cardoso JMB, Cardoso MH. Predicting postoperative atrial fibrillation after myocardial revascularization without cardiopulmonary bypass: A retrospective cohort study. J Card Surg. 2019 Jul;34(7):577-582. doi: 10.1111/jocs.14088. Epub 2019 Jun 18. PMID 31212388
- [Result] Kirchhof P, Breithardt G, Camm AJ, Crijns HJ, Kuck KH, Vardas P, Wegscheider K. Improving outcomes in patients with atrial fibrillation: rationale and design of the Early treatment of Atrial fibrillation for Stroke prevention Trial. Am Heart J. 2013 Sep;166(3):442-8. doi: 10.1016/j.ahj.2013.05.015. Epub 2013 Jul 30. PMID 24016492
- [Result] Hanna P, Buch E, Stavrakis S, Meyer C, Tompkins JD, Ardell JL, Shivkumar K. Neuroscientific therapies for atrial fibrillation. Cardiovasc Res. 2021 Jun 16;117(7):1732-1745. doi: 10.1093/cvr/cvab172. PMID 33989382
- [Result] Nso N, Bookani KR, Metzl M, Radparvar F. Role of inflammation in atrial fibrillation: A comprehensive review of current knowledge. J Arrhythm. 2020 Dec 23;37(1):1-10. doi: 10.1002/joa3.12473. eCollection 2021 Feb. PMID 33664879
- [Result] Connors CW, Craig WY, Buchanan SA, Poltak JM, Gagnon JB, Curry CS. Efficacy and Efficiency of Perioperative Stellate Ganglion Blocks in Cardiac Surgery: A Pilot Study. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):e28-e30. doi: 10.1053/j.jvca.2017.10.025. Epub 2017 Oct 20. No abstract available. PMID 29162313
- [Result] Leftheriotis D, Flevari P, Kossyvakis C, Katsaras D, Batistaki C, Arvaniti C, Giannopoulos G, Deftereos S, Kostopanagiotou G, Lekakis J. Acute effects of unilateral temporary stellate ganglion block on human atrial electrophysiological properties and atrial fibrillation inducibility. Heart Rhythm. 2016 Nov;13(11):2111-2117. doi: 10.1016/j.hrthm.2016.06.025. Epub 2016 Jun 21. PMID 27353237
- [Result] Puente de la Vega Costa K, Gomez Perez MA, Roqueta C, Fischer L. Effects on hemodynamic variables and echocardiographic parameters after a stellate ganglion block in 15 healthy volunteers. Auton Neurosci. 2016 May;197:46-55. doi: 10.1016/j.autneu.2016.04.002. Epub 2016 Apr 16. PMID 27143533